CLINICAL TRIAL: NCT00915681
Title: A Phase II Multi-Center Open-Label Clinical Trial to Assess the Prevention of Liver Transplantation and/or Death Among Subjects Treated With Intravenous Silibinin (Legalon® SIL) for Amatoxin Induced Hepatic Failure
Brief Title: Intravenous Milk Thistle (Silibinin-Legalon) for Hepatic Failure Induced by Amatoxin/Amanita Mushroom Poisoning
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Mylan Specialty, LP (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB16A1.07
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-01

CONDITIONS: Amatoxin Poisoning; Amanita Poisoning; Mushroom Poisoning; Liver Failure
Keywords: amatoxin; amanita; mushroom poisoning; hepatic failure; milk thistle; Silibinin; Legalon
MeSH Terms: conditions — Mushroom Poisoning; Liver Failure | interventions — Silybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Legalon SIL (Experimental): Silibinin: loading dose of one hour infusion of 5 mg/kg, followed by 20 mg/kg/day infused continuously via pump
  Interventions: Drug: Silibinin

INTERVENTIONS:
Drug: Silibinin — 20 mg/kg continuous IV is over 24 hours
  Other Names: Legalon SIL

SUMMARY:
Legalon® SIL will be administered to patients with amatoxin poisoning diagnosed by history, gastrointestinal symptoms, elevated liver enzymes, and/or diagnostic assay (should one become available). Patients may or may not also demonstrate abnormalities in bilirubin and/or creatinine. Treatment consists of a 5 mg/kg loading dose followed by 20 mg/kg/day via continuous infusion. The treating physician is expected to administer supportive therapy of his/her choosing but consistent with best practices. Legalon® SIL will be stopped when coagulopathy is no longer present, and when liver function tests have returned significantly towards the normal range. Patients will be followed 7-14 days after the end of Legalon® SIL therapy with follow up lab studies.

DETAILED DESCRIPTION:
Patients with suspected amatoxin poisoning are reviewed for enrollment in the study by contacting the Legalon SIL study hotline (866) 520-4412.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent(s) for clinical trial participation (due to the potential critical status of the subject upon presentation, consent may need to be obtained from Legally Authorized Representative (LAR) per sites consenting policy and ICH/GCP guidance) Signed Informed Consent for Clinical Trial participation
2. History of eating foraged mushrooms
3. Gastrointestinal symptoms suggestive of amatoxin poisoning (cramping abdominal pain, nausea, vomiting, and / or watery diarrhea) usually 24-48 hours after of mushroom ingestion
4. Liver function tests suggestive of amatoxin poisoning: AST or ALT above the institutions upper limit of normal after mushroom ingestion

Exclusion criteria:

1. Evidence of significant medical illness or any other abnormal laboratory finding that, in the Investigator's judgment, will substantially increase the risk associated with the subject's participation in, and completion of the study or could preclude the evaluation of the subject's response.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-11-10 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wallis Marsh, MD, Principal Investigator — WVU
Locations (2):
- United States (2):
  - Recruitment Hot Line for the United States, Somerset, New Jersey
  - Mylan Specialty LLP, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 148 screened, 102 treated FPI: 10-Nov-2009, LPO: 10-Apr-2020
Groups:
- Legalon SIL: Silibinin: loading dose of one hour infusion of 5 mg/kg, followed by 20 mg/kg/day infused continuously via pump
  Silibinin: 20 mg/kg/day IV
Period: Overall Study
Arm/Group | Legalon SIL
Started | 148
Completed | 102
Not Completed | 46
Not completed — Screening failures | 46

BASELINE CHARACTERISTICS:
Population: Study was terminated, no analysis performed as data are unavailable for most patients.
Arm/Group | Legalon SIL
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants] — Population: data are unavailable for 31 patients out of the 102 treated patients
  Participants
    number analyzed (Participants) | 71
    <=18 years | 4
    Between 18 and 65 years | 41
    >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: data are unavailable for 31 patients out of the 102 treated patients
  years
    number analyzed (Participants) | 71
    (all) | 54.9 (19.89)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: data are unavailable for 31 patients out of the 102 treated patients
  Participants
    number analyzed (Participants) | 71
    Female | 37
    Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: data are unavailable for 31 patients out of the 102 treated patients
  participants
    United States: number analyzed (Participants) | 71
    United States | 71

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Percentage of Subjects Treated Under This Clinical Trial Without Morbidity (Liver Transplantation) and or Mortality (Death).
Description: Study was terminated, no analysis performed as data are unavailable for most patients
Time Frame: not applicable as no analysis was performed
Population: The data is determined to be unreliable and this has been communicated to FDA and the IRB/EC; Therefore the study data cannot be analyzed and summarized to be reported except for the basic information.
Arm/Group | Legalon SIL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 10 days
Arm/Group | Legalon SIL
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Mylan is allowed to require modifications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT00915681/Prot_SAP_000.pdf